CLINICAL TRIAL: NCT06227429
Title: A Prospective, Non-interventional, Post-Marketing Study to Describe Outcome of Nitisinone Treatment in Hereditary Tyrosinemia Type 1 (HT-1) Patients in Routine Clinical Care in China
Brief Title: A Non-interventional, Post-Marketing Study to Describe Outcome of Nitisinone Treatment in HT-1 Patients
Status: Withdrawn | Type: Observational
Why Stopped: No patients were prescribed to the study treatment due to the generic treatment being available.
Sponsor: Swedish Orphan Biovitrum (Industry)
Responsible Party: Sponsor
Other Study IDs: Sobi.NTBC-008
Record Dates: First submitted 2023-12-19; First posted 2024-01-26 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Hereditary Tyrosinemia, Type I
Keywords: rare diseases; fumarylacetoacetate hydrolase (FAH) deficiency; liver failure; drug treatment; nitisinone; observational research; phase IV; China; pediatric patient
MeSH Terms: conditions — Tyrosinemias; Rare Diseases; Fanconi Anemia; Liver Failure | interventions — nitisinone

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Full Analysis Set (FAS): The Full Analysis Set (FAS) will include all patients with a confirmed HT-1 diagnosis on Nitisinone treatment in routine clinical care, who provide signed informed consent. Patients must be either on treatment with Nitisinone at study entry or they must have been prescribed Nitisinone at enrollment. No specific exclusion criteria from the analysis set will be applied. The FAS will be used for all analyses.
  Interventions: Drug: Nitisinone

INTERVENTIONS:
Drug: Nitisinone — According to prescription
  Other Names: Orfadin®

SUMMARY:
This is a prospective, non-interventional, non-comparative, multicenter study to collect data on HT-1 patients in China treated with Nitisinone in a routine clinical setting. No tests or examinations are mandated in the study.

DETAILED DESCRIPTION:
This is a prospective, non-interventional, non-comparative, multicenter study to collect data on HT-1 patients in China treated with Nitisinone in a routine clinical setting. No tests or examinations are mandated in the study, though the expectation is that most of the tests and examinations listed in the protocol will be performed in the context of routine clinical care and relevant data will be captured. At enrollment, data on patient treatment, medical and surgical history together with other patient characteristics will be captured.Patients enrolled in the study will be followed for at least 1 year and for a maximum of 3.5 years.

The study aims to enroll at least 15 HT-1 patients aged 0-18 years. If adult patients are enrolled the study population will be larger as all eligible patients will be invited to participate. However, the enrollment will close when the target of 15 patients aged 0-18 years has been reached.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a confirmed diagnosis of HT-1 treated with, or at enrollment prescribed, Nitisinone treatment (product manufactured by Sobi) in a routine clinical care setting. The decision to initiate treatment shall be made by the treating physician independently from the decision to include the patient in the study.
2. Signed and dated informed consent provided by the patient, or the patient's legally authorized representative(s) for patients under the legal age, should be obtained before any study-related activities are undertaken. Assent should be obtained from pediatric patients according to local regulations

Exclusion Criteria:

1. Enrollment in a concurrent clinical interventional study, or intake of an Investigational Medicinal Product (IMP), within three months prior to inclusion in this study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Investigators at selected sites in China will attempt to consecutively enroll all eligible patients who present for a routine clinical visit.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Occurrence of hepatic, renal or hematological adverse events (AEs) or death | Data will be collected for all routine visits completed during the study period which is at least 12 months but no more than 3.5 years.
  Number and percent of patients with occurrence and number of occurrences per 100 patient years.

SECONDARY OUTCOMES:
Occurrence of death | Data will be collected for all routine visits completed during the study period which is at least 12 months but no more than 3.5 years.
  Number and percent of patients with occurrence and number of occurrences per 100 patient years.
Occurrence of liver transplantation | Data will be collected for all routine visits completed during the study period which is at least 12 months but no more than 3.5 years.
  Number and percent of patients with occurrence and number of occurrences per 100 patient years.
Occurrence of hepatic malignancy | Data will be collected for all routine visits completed during the study period which is at least 12 months but no more than 3.5 years.
  Number and percent of patients with occurrence and number of occurrences per 100 patient years.
Occurrence of other (non-hepatic) malignancies | Data will be collected for all routine visits completed during the study period which is at least 12 months but no more than 3.5 years.
  Number and percent of patients with occurrence and number of occurrences per 100 patient years.
Occurrence of ophthalmic events | Data will be collected for all routine visits completed during the study period which is at least 12 months but no more than 3.5 years.
  Number and percent of patients with occurrence and number of occurrences per 100 patient years.
Occurrence of neurological events | Data will be collected for all routine visits completed during the study period which is at least 12 months but no more than 3.5 years.
  Number and percent of patients with occurrence and number of occurrences per 100 patient years.
Occurrence of cognitive, developmental function AEs | Data will be collected for all routine visits completed during the study period which is at least 12 months but no more than 3.5 years.
  Cognitive, developmental function AEs will be recorded in the eCRF.
Occurrence of any reportable AEs | Data will be collected for all routine visits completed during the study period which is at least 12 months but no more than 3.5 years.
  Number and percent of patients with occurrence and number of occurrences per 100 patient years.
  Reportable AEs are defined as:
  * All Serious Adverse Events (SAEs) irrespective of causality with Nitisinone
  * Non-serious Adverse Events (AEs) assessed as causally related to treatment with Nitisinone
  * All Adverse Events leading to subject discontinuation from the study
Treatment and diet compliance | Data will be collected for all routine visits completed during the study period which is at least 12 months but no more than 3.5 years.
  Rated from 1 ("very good") to 4 ("very poor") and "unknown". Number and percent of patients in each group.
Extent of exposure | Data will be collected for all routine visits completed during the study period which is at least 12 months but no more than 3.5 years.
  Extent of exposure as measured by:
  * Prescribed daily dose of Nitisinone
  * Changes in prescribed doses of Nitisinone
Extent of Exposure | Data will be collected for all routine visits completed during the study period which is at least 12 months but no more than 3.5 years.
  Extent of exposure as measured by:
  * Nitisinone trough concentrations in dried blood spot
  * Nitisinone trough concentrations in serum or plasma (depending on method)
Laboratory investigations - Blood Coagulation (1) | Data will be collected for all routine visits completed during the study period which is at least 12 months but no more than 3.5 years.
  Mean, median, standard deviation, minimum, and maximum time for ad-hoc specified age groups will be calculated for:
  • Prothrombin time (International Normalized Ratio)
Laboratory investigations - Blood Coagulation (2) | Data will be collected for all routine visits completed during the study period which is at least 12 months but no more than 3.5 years.
  Mean, median, standard deviation, minimum, and maximum time for ad-hoc specified age groups will be calculated for:
  • Partial thromboplastin time (milliseconds)
Laboratory investigations - Blood Coagulation (3) | Data will be collected for all routine visits completed during the study period which is at least 12 months but no more than 3.5 years.
  Mean, median, standard deviation, minimum, and maximum time for ad-hoc specified age groups will be calculated for:
  • Activated partial thromboplastin time (seconds per ration)
Laboratory investigations - Blood Chemistry (1) | Data will be collected for all routine visits completed during the study period which is at least 12 months but no more than 3.5 years.
  Mean, median, standard deviation, minimum, and maximum concentration for ad-hoc specified age groups will be calculated for blood concentrations of:
  * Tyrosine (µmol/L)
  * Phenylalanine (µmol/L)
  * Succinylacetone (µmol/L)
  * Creatinine (µmol/L)
  * Aspartate transaminase (µmol/L)
  * Serum bilirubin (µmol/L)
Laboratory investigations - Blood Chemistry (2) | Data will be collected for all routine visits completed during the study period which is at least 12 months but no more than 3.5 years.
  Mean, median, standard deviation, minimum, and maximum concentration for ad-hoc specified age groups will be calculated for blood concentrations of:
  • Alpha-fetoprotein (ng/mL)
Laboratory investigations - Blood Chemistry (3) | Data will be collected for all routine visits completed during the study period which is at least 12 months but no more than 3.5 years.
  Mean, median, standard deviation, minimum, and maximum concentration for ad-hoc specified age groups will be calculated for blood concentrations of:
  * Alanine transaminase (international units per liter)
  * Alkaline phosphatase (international units per liter)
  * Gamma-glutamyl transferase (international units per liter)
Laboratory investigations - Blood Chemistry (4) | Data will be collected for all routine visits completed during the study period which is at least 12 months but no more than 3.5 years.
  Mean, median, standard deviation, minimum, and maximum concentration for ad-hoc specified age groups will be calculated for blood concentrations of:
  • Albumin (g/L)
Overall clinical condition as assessed by the investigator | Data will be collected for all routine visits completed during the study period which is at least 12 months but no more than 3.5 years.
  Overall clinical condition will be assessed by the investigator on a 4-point scale; normal, mildly ill, moderately ill, markedly ill. Number and percent of patients in each group.
Ophthalmic status as assessed by the investigator | Data will be collected for all routine visits completed during the study period which is at least 12 months but no more than 3.5 years.
  As assessed by the investigator ("yes, normal", "no, not normal", and "unknown"). Number and percent of patients in each group.
Neurocognitive/developmental status as assessed by the investigator | Data will be collected for all routine visits completed during the study period which is at least 12 months but no more than 3.5 years.
  As assessed by the investigator ("yes, normal", "no, not normal", and "unknown"). Number and percent of patients in each group.

CONTACTS AND LOCATIONS:
Overall Officials: Ioannis Kottakis, MD, PhD, Study Director — Swedish Orphan Biovitrum; Xiaoping Luo, MD, PhD, Principal Investigator — Tongji Hospital, Tongji Medical College of Huazhong University of Science & Technology
Locations (4):
- China (4):
  - Swedish Orphan Biovitrum Research Site, Beijing
  - Swedish Orphan Biovitrum Research Site, Chongqing
  - Swedish Orphan Biovitrum Research Site, Hefei
  - Swedish Orphan Biovitrum Research Site, Wuhan

IPD SHARING:
Plan to Share IPD: Yes
According to Sobi's data sharing policy Sobi may share anonymized clinical study data with qualified researchers. Sobi commits to sharing clinical study data on participant level and summary data for medicines and indications approved by the European Medicines Agency (EMA) and/or the Food and Drug Administration (FDA). Data access will be granted in response to qualified research requests. All requests are evaluated by a cross functional panel of experts within Sobi.
Time Frame: Evaluated on a case by case basis
Access Criteria: A decision on data sharing will be based on the following:
  * The scientific merit of the proposal - i.e. the proposal should be scientifically sound, ethical, and have the potential to contribute to the advancement of public health.
  * The feasibility of the research proposal - i.e. the requesting research team must be scientifically qualified and have the resources to conduct the proposed project.
  * Maintenance of personal integrity - i.e. Sobi will not consider sharing individual data if there is a risk of re-identification of individuals despite a proper anonymisation. Moreover, the patients' informed consent will always be respected. Sobi reserves the right to reject the proposal if the anonymisation process will render unusable data.
  * Publication of results - the applicants should commit to submit their findings to a peer-reviewed scientific journal, alternatively to present the results at a congress (poster or similar), regardless of the research outcome
URL: https://www.sobi.com/en/policies